CLINICAL TRIAL: NCT02012686
Title: The Effect of Transcutaneous Electrical Nerve Stimulation for Reduction of Posterior Neck Pain After Thyroidectomy
Brief Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Posterior Neck Pain After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Cholhee Park, clinical assisted professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20131127
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-05

CONDITIONS: Thyroid Cancer; Neck Pain
Keywords: transcutaneous electric nerve stimulation; thyroidectomy; neck pain; pain management
MeSH Terms: conditions — Thyroid Neoplasms; Neck Pain; Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): numerical rating scale of TENS non-applied group
- TENS group (Active Comparator): numerical rating scale of TENS applied group
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — transcutaneous electric nerve stimulation frequency of 100 Hz pulse duration of 200 µs wih stimulation intensity of feeling strong but non-painful paresthesia in the upper trapezius
  Other Names: LT1061 (Shenzhen Dongdixin Technology, Shenzhen, China)
  Arms: TENS group

SUMMARY:
The purpose of tihs study is to determine whether transcutaneous electric nerve stimulation (TENS) during thyroidectomy is effective in the reduction of posterior neck pain after thyroidectomy.

DETAILED DESCRIPTION:
Thyroidectomy is performed in supine position with the neck fully extended. After thyroidectomy, 80 percent of patients experience posterior neck pain as well as the incision site pain. The posterior neck pain is thought to be due to hyperextension is continued during an average of 90 minutes of surgery. Non-steroidal anti-inflammatory agents or opioids are administrated to reduce the pain, but the pain still remained.

TENS is simple, non-invasive analgesic technique that is used extensively to reduce acute and chronic pain. TENS has beneficial effect for the reduction of postoperative pain. The conventional way of administering TENS is to use electric characteristics that selectively activate large diameter Aβ fiber mediating touch perception without activating smaller diameter Aδ and C fiber.

In this study, TENS during thyroidectomy in posterior neck pain will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing open total thyroidectomy under general anesthesia
* American Society of Anesthesiology physical status I or II

Exclusion Criteria:

* American Society of Anesthesiology physical status III or IV
* History of headache or neck pain within six months
* Past history of herniated cervical disc, cervical foraminal stenosis, ossification of posterior longitudinal ligament

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Woo Han, M.D.,ph.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, Gangnam Severance Hospital, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, 211 Eonju-ro, Gangnam-gu, Seoul 135-720, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Gangnam Severance Hospital, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- TENS Group: numerical rating scale of TENS applied group
  TENS: transcutaneous electric nerve stimulation
Period: Overall Study
Arm/Group | Control Group | TENS Group
Started | 50 | 50
Completed | 50 | 48
Not Completed | 0 | 2
Not completed — muscle contraction | 0 | 1
Not completed — electrocardiography monitoring noise | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | TENS Group | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10) | 44 (9) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 50 | 48 | 98
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23 (3) | 23 (3) | 23 (3)
Neck extension time [Mean (Standard Deviation); unit: minutes] — neck extension time: neck extension position time for thyroidectomy (Just after general anesthesia, the neck of patient was extended. The position was kept before awakening)
  minutes | 80 (25) | 81 (31) | 80 (28)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale of Posterior Neck Pain 0.5 Hours After Thyroidectomy
Description: numerical rating scale from 0 - 10. where 0 indicates no pain and 10 indicates the worst pain imaginable
Time Frame: 0.5 hours after thyroidectomy
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Control Group | TENS Group
Number analyzed (Participants) | 50 | 48
scores on a scale
  Inter-Quatile Range | 3.5 [1 to 5] | 0 [0 to 2]
  Full Range | 3.5 [0 to 10] | 0 [0 to 6]

2. Primary Outcome: Numerical Rating Scale of Posterior Neck Pain 6 Hours After Thyroidectomy
Description: numerical rating scale from 0 - 10. where 0 indicates no pain and 10 indicates the worst pain imaginable
Time Frame: 6 hours after thyroidectomy
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Control Group | TENS Group
Number analyzed (Participants) | 50 | 48
scores on a scale
  Inter-Quatile Range | 4 [3 to 5] | 2 [0 to 4]
  Full Range | 4 [0 to 8] | 2 [0 to 8]

3. Primary Outcome: Numerical Rating Scale of Posterior Neck Pain 24 Hours After Thyroidectomy
Description: numerical rating scale from 0 - 10. where 0 indicates no pain and 10 indicates the worst pain imaginable
Time Frame: 24 hours after thyroidectomy
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Control Group | TENS Group
Number analyzed (Participants) | 50 | 48
scores on a scale
  Inter-Quatile Range | 3 [2 to 4] | 1 [0 to 3]
  Full Range | 3 [0 to 6] | 1 [0 to 5]

4. Primary Outcome: Numerical Rating Scale of Posterior Neck Pain 48 Hours After Thyroidectomy
Description: numerical rating scale from 0 - 10. where 0 indicates no pain and 10 indicates the worst pain imaginable
Time Frame: 48 hours after thyroidectomy
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Control Group | TENS Group
Number analyzed (Participants) | 50 | 48
scores on a scale
  Inter-Quatile Range | 2 [0 to 4] | 0 [0 to 2]
  Full Range | 2 [0 to 5] | 0 [0 to 6]

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Control Group | TENS Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No